CLINICAL TRIAL: NCT04187820
Title: Effect of Acupuncture on Crohn's Disease Via the Regulation of Trp-kyn Metabolism in Brain-gut Axis
Brief Title: Effect of Acupuncture on Mild to Moderate Active Crohn's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Collaborators: Fudan University (Other); Shanghai University of Traditional Chinese Medicine (Other); Shanghai Jiao Tong University School of Medicine (Other); Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYS2019-01
Record Dates: First submitted 2019-12-01; First posted 2019-12-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Intestinal Disorder; Inflammatory Bowel Diseases; Crohn Disease
Keywords: acupuncture; Crohn's disease
MeSH Terms: conditions — Intestinal Diseases; Inflammatory Bowel Diseases; Crohn Disease | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture group (Experimental): Participants receiving acupuncture and mild moxibustion.
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — Patients receiving acupuncture and mild moxibustion, whom were treated 3 times per week for 12 weeks and followed up for 36 weeks. CV12 and Bilateral ST37, SP6, SP4, LR3, KI3, LI4 and LI11 were selected for acupuncture and bilateral ST25 and ST36 were selected for moxibustion. In the acupuncture group, Hwato acupuncture device was used to blind the subjects, and had the deqi sensation. The surface temperature of acupoints was maintained at 43℃± 1℃ for moxibustIon.

SUMMARY:
To observe the clinical effect of acupuncture on Crohn's disease (CD) and its influence on brain function activity and the TRY-KYN metabolism level, and to screen the brain image markers of acupuncture on CD

DETAILED DESCRIPTION:
1. Effect of acupuncture on symptoms of CD
2. Effect of acupuncture on brain functional activity of CD
3. Effect of acupuncture on intestinal and plasma TRP-KYN metabolism level of CD
4. Screen the brain image markers of acupuncture in the treatment of CD

ELIGIBILITY:
Inclusion Criteria:

1. aged 16-70;
2. patients with mild or moderate active disease (150 ≤ CDAI < 450);
3. patients who are not responsive, intolerant, dependent or refused to use at least mesalazine, glucocorticoid, immunomodulator (azathioprine, methotrexate), anti TNF alpha preparation;
4. patients were not taking medication or were only taking one or more of the following drugs: [prednisone ≤15mg/d, azathioprine (≤1mg/kg/d), methotrexate (≤15mg/w) or mesalazine (≤4g/d)] and prednisone was used for at least 1 month, while azathioprine, methotrexate or mesalazine was used for at least 3 months;
5. those who did not use anti-TNF alpha and other agents within 3 months before entering the study;
6. those who have never experienced acupuncture;
7. patients signing informed consent.

Exclusion Criteria:

1. patients who are recently pregnant or in pregnancy or lactation;
2. patients with serious organic diseases;
3. patients diagnosed as psychosis;
4. patients who take antibiotics, probiotics, traditional Chinese medicine and other drugs at the same time, or who suffer from multiple diseases and need to take other drugs for a long time, and may affect the observation of the efficacy of this trial;
5. severe skin diseases (such as erythema nodosum, pyoderma gangrenosum, etc.), eye diseases (such as iritis, uveitis, etc.), thromboembolic diseases and other serious extraintestinal manifestations;
6. there are serious intestinal fistula, abdominal abscess, intestinal stenosis and obstruction, perianal abscess, gastrointestinal hemorrhage, intestinal perforation and other complications;
7. patients with short bowel syndrome who have undergone abdominal or gastrointestinal surgery in the past half a year;
8. there are skin diseases or defects in the selected area of acupuncture and moxibustion that cannot be performed.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | Week 12
  Crohn's disease activity index （CDAI）less than 150 and decreased more than 70

SECONDARY OUTCOMES:
Clinical remission | Week 24, 36 and 48
  Crohn's disease activity index （CDAI） less than 150 and decreased more than 70
Clinical response | Week 12, 24, 36 and 48
  Crohn's disease activity index （CDAI） decreased more than 70
Crohn's disease activity index （CDAI）score | Week 12, 24, 36 and 48
  The mean change in CDAI from baseline. The higher the score, the worse the condition. Greater than 0, no upper limit.
laboratory test | Week 12, 24, 36 and 48
  serum C-reactive protein (CRP) level
laboratory test | Week 12, 24, 36 and 48
  Erythrocyte sedimentation rate (ESR)
laboratory test | Week 12, 24, 36 and 48
  Platelet count
Inflammatory bowel disease questionnaire (IBDQ) | Week 12 and 24
  The mean change in IBDQ from baseline. The higher the score, the worse the condition.The score is range from 32 to 224.
Crohn's disease endoscopic index of severity (CDEIS) | Week 48
  The mean change in CDEIS from baseline
Hospital anxiety and depression scale (HADS) | Week 12 and 24
  The mean change in HADS from baseline. The higher the score, the more serious the disease. The depression and anxiety score is range from 0 to 21.
The proportion of recurrences | Week 48
  Defined as CDAI > 150 and increase ≥ 70 points or need to adjust drug to control disease condition.
Brain functional and structural changes | Week 12
  measured by functional MRI
Plasma and intestinal TRP-KYN metabolism level | Week 12
  Plasma and intestinal Indoleamine2,3dioxygenase 1 （IDO1）level
Plasma and intestinal TRP-KYN metabolism level | Week 12
  Plasma and intestinal Tryptophan (TRP) level
Plasma and intestinal TRP-KYN metabolism level | Week 12
  Plasma and intestinal kynurenine （KYN）level
Plasma and intestinal TRP-KYN metabolism level | Week 12
  Plasma and intestinal kynurenic acid （KYNA） level
Plasma and intestinal TRP-KYN metabolism level | Week 12
  Plasma and intestinal quinolinic acid (QUIN) level
Plasma and intestinal TRP-KYN metabolism level | Week 12
  Plasma and intestinal IFN-gamma level
Plasma and intestinal TRP-KYN metabolism level | Week 12
  Plasma and intestinal IL-1beta level
Plasma and intestinal TRP-KYN metabolism level | Week 12
  Plasma and intestinal IL-18 level

OTHER OUTCOMES:
Analysis of intestinal microbes | Week 12
  Application of 16S sequencing to analyze the gut microbial composition, structure and diversity of patients.
Analysis of the association between gut microbes, brain imaging and behavior | Week 12
  The pearson correlation and linear regression models were applied to establish the association between gut microbes, brain function and structure and behavior in an attempt to explore the relationship between the gut microbe-gut-brain axis in patients with active CD.
Acupuncture efficacy prediction | Week 48
  Deep learning algorithms such as artificial neural networks and support vector machines were applied to construct and validate an acupuncture efficacy prediction model based on MRI changes in high and low response patients in the acupuncture group, and to screen brain neuroimaging markers that predict the effective relief of CD disease activity by acupuncture.
Disease activity prediction | Week 0
  Differences in brain structure and functional activity between active CD patients and remitting CD patients as well as healthy subjects are measured, and deep learning algorithms such as artificial neural networks and support vector machines are applied to construct and validate disease diagnostic models and screen brain imaging markers that predict CD disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Huangan Wu, MD, PhD, Study Chair — Shanghai Research Institute of Acupuncture and Meridian
Locations (2):
- China (2):
  - Shanghai Research Institute of Acupuncture and Meridian, Shanghai, Shanghai Municipality
  - Guona Li, Shanghai

IPD SHARING:
Plan to Share IPD: No